CLINICAL TRIAL: NCT03410979
Title: A 2-part, Randomized, Double-blind, Placebo-controlled, Sequential Group, Dose-escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG2737 in Healthy Male Subjects
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of GLPG2737 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG2737-CL-101; 2016-003626-17 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLPG2737 single dose (Experimental): Single doses of GLPG2737 oral suspension at up to 5 dose levels in ascending order
  Interventions: Drug: GLPG2737 single dose
- Placebo single dose (Placebo Comparator): Single doses of Placebo oral suspension
  Interventions: Drug: Placebo single dose
- GLP2737 multiple dose (Experimental): Multiple doses of GLPG2737 oral suspension at up to 3 dose levels in ascending order
  Interventions: Drug: GLPG2737 multiple dose
- GLPG2737 multiple dose (Placebo Comparator): Multiple doses of Placebo oral suspension
  Interventions: Drug: GLPG2737 multiple dose

INTERVENTIONS:
Drug: GLPG2737 single dose — GLPG2737 oral suspension, single ascending doses
  Arms: GLPG2737 single dose
Drug: Placebo single dose — Placebo, oral suspension.
  Arms: Placebo single dose
Drug: GLPG2737 multiple dose — GLPG2737 oral suspension, multiple ascending doses, daily for 14 days.
  Arms: GLP2737 multiple dose
Drug: GLPG2737 multiple dose — Placebo, oral suspension, daily for 14 days
  Arms: GLPG2737 multiple dose

SUMMARY:
This study is a first-in-human (FIH), Phase I, single center, randomized, double-blind, placebo-controlled, sequential group study in healthy male subjects to assess the safety, tolerability and PK of single ascending oral doses of GLPG2737 and multiple ascending oral doses of GLPG2737 administered for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18-50 years of age, inclusive, on the date of signing the Informed Consent Form (ICF).
2. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and clinical safety laboratory tests prior to the initial study drug administration.

   Clinical safety laboratory test results must be within the laboratory reference ranges for males or test results that are outside the reference ranges for males need to be considered non clinically significant in the opinion of the investigator. One retest is allowed if deemed appropriate by the investigator.
3. Liver function tests must meet the following criteria:

   1. aspartate aminotransferase (AST), ALT or alkaline phosphatase (ALP) <1.2x the upper limit of normal (ULN)
   2. Bilirubin not greater than ULN, however documented Gilbert's syndrome is acceptable. One retest is allowed if deemed appropriate by the investigator.
4. Subject's screening ECG is considered normal or abnormal but clinically non-significant. QTcF must not exceed 450 msec. First degree heart block will not be considered as a significant abnormality.
5. Forced expiratory volume in 1 second (FEV1) ≥ 80% of predicted normal for age, gender and height at screening.
6. Discontinuation of all medications (including over-the-counter and/or prescription medication, dietary supplements, nutraceuticals, vitamins and/or herbal supplements) except occasional paracetamol (maximum dose of 2 g/day and maximum of 10 g/2 weeks) at least 2 weeks prior to the first study drug administration.
7. Negative drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) prior to dosing.
8. Able and willing to comply with the prohibitions and restrictions as described in the protocol and with the contraceptive requirements as described in the protocol.
9. Able and willing to sign the ICF as approved by the IEC, prior to any screening evaluations.

Exclusion Criteria:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A.
3. History of or a current immunosuppressive condition (e.g., human immunodeficiency virus [HIV] infection type 1 and 2).
4. Clinically significant illness in the 3 months before screening.
5. Presence or having sequelae of gastrointestinal, liver (except for Gilbert's syndrome), kidney (creatinine clearance ≤ 80 mL/min using the Cockcroft-Gault formula: if calculated result ≤ 80 mL/min, a 24 hour urine collection to determine actual value can be done) or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
6. History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated and with no evidence of recurrence).
7. Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months of 5-half-lives of the drug (whichever is longer) before the initial drug administration.
8. Active drug or alcohol abuse (an average intake of more than 21 glasses of wine or beer or equivalent/week) within 2 years prior to screening.
9. Participation in a drug, drug/device or biologic investigational research study within 12 weeks or 5 half-lives of the investigational drug, if the half-life is known (whichever is longer) prior to screening.
10. Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in the proportion of subjects with adverse events | Between screening and 14 days (SAD part) and 15 days (MAD part) after the last dose
  To assess safety and tolerability of single and multiple ascending doses with GLPG2737 versus placebo in healthy subjects.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG2737 | Between Day 1 predose and 5 days after the last dose
  To characterize pharmacokinetics of GLPG2737 and its metabolites after single and multiple oral doses in healthy subjects
Time of occurrence of Cmax for GLPG2737 (tmax) | Between Day 1 predose and 5 days after the last dose
  To characterize pharmacokinetics of GLPG2737 and its metabolites after single and multiple oral doses in healthy subjects
Area under the plasma concentration-time curve (AUC0-t) of GLPG2737 | Between Day 1 predose and 5 days after the last dose
  To characterize pharmacokinetics of GLPG2737 and its metabolites after single and multiple oral doses in healthy subjects
Ratio of 4-beta-hydroxycholesterol/cholesterol in plasma after multiple oral doses in healthy subjects | Day 1 predose and Day 14
  To explore the potential of CYP3A4 interaction with GLPG2737

CONTACTS AND LOCATIONS:
Overall Officials: Chris Brearley, BM, MRCP, MFPM, Study Director — Galapagos NV
Locations (1):
- PRA-EDS, Groningen, Netherlands